CLINICAL TRIAL: NCT05852444
Title: Comparison of Postoperative Pain After Using Passive Ultra Sonic Activation (PUA) and Manual Dynamic Agitation (MDA) During Root Canal Treatment
Brief Title: Evaluation of Post Operative Pain After Ultrasonic Activation and Manual Dynamic Agitation As Final Irrigation Protocols During Root Canal Treatment
Acronym: Ultra X
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Ahmed Abdullah, Registrar Operative Dentistry and Endodontics, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ultrasonic Activation
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants to be divided into 2 different groups randomly, and intervention protocol to be performed as per group designation
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants of the study and outcomes assessor would not know the details of groups, and only the investigator and care provider would be aware of that, as they cannot be blinded due to the nature of this study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Manual Dynamic Agitation Group: Irrigation in this group shall be done using a master gutta percha cone during root canal therapy
  Interventions: Device: Manual Dynamic Agitation
- Group B (Experimental): Passive Ultrasonic Activation Group: In this group, final activation during endodontic therapy shall be done using an ultrasonic activation device (Ultra X)
  Interventions: Device: Passive Ultrasonic Activation

INTERVENTIONS:
Device: Passive Ultrasonic Activation — Agitation of root canal irrigation solution with an ultrasonic activation device (Ultra X).
  Arms: Group B
Device: Manual Dynamic Agitation — Agitation of root canal irrigation solution with master gutta percha cone
  Arms: Group A

SUMMARY:
The study analyzes the difference in post operative pain after root canal therapy, after using different activation protocols and devices. The subjects are divided into 2 groups and a different activation protocol is used in each group. In one group, final activation of irrigating agent during root canal therapy is done with an ultrasonic activation device, and in the other group, manual dynamic agitation is done using master gutta percha cone. The Post operative pain is then compared at 8, 24,and 48 hour intervals

DETAILED DESCRIPTION:
Root canal therapy is a procedure in which inflamed pulp tissue and microorganisms are removed from root canals and pulp chamber, in order to eradicate infection and symptoms. Irrigation is a crucial step of an endodontic therapy and different methods and protocols are used to enhance the efficacy of irrigation. Ultrasonic activation of root canal irrigation agent is one of the effective methods that enhance the outcomes and success rate of endo therapies. It removes the smear layer, bacterial biofilms and debris by acoustic streaming and agitating the irrigant inside root canals. Similarly, a conventional method of agitation (manual dynamic agitation) also play an important role in endodontic therapy, particularly by improving the delivery of irrigation agent to the apex of a root canal. The later method involves agitation of irrigant with master gutta percha cone with continuous to and fro strokes manually.

In this study, the efficacy of both the different irrigation protocols will be compared and assessed based on post-operative pain, measured by Visual Analog Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unremarkable/ noncontributory medical history
2. Healthy persons between the ages of 18 and 60 years
3. Maxillary and mandibular molar teeth diagnosed with symptomatic irreversible pulpitis.
4. Patients not having taken any medication for 6 hours before treatment
5. No allergies to the drugs or dental material being used in the treatment

Exclusion Criteria:

1. Patients who had taken analgesics on anti-inflammatory drugs within the last 12 hours
2. Pregnant women and patients with immunocompromised health state
3. Patients having severe malocclusion associated with traumatic occlusion
4. Teeth with calcified canals
5. Teeth with periapical radiolucency
6. Teeth with root resorption
7. Teeth previously undergone root canal treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
Post Operative pain assessed by VAS after endodontic therapy | 1 week
  comparative evaluation of post operative pain after using different irrigation devices, using VAS (Visual Analog Scale). It is drawn as a straight line of 10 inches and marked in numbers which show intensity of pain, from 0-10, with 0 being no pain at all to10 being the worst pain imaginable. In detail, it is a scale which shows pain intensity in ascending order and can also be used to analyze the intensity of pain experienced by the patient.
  0: No pain at all 1-3: mild pain 4-6: moderate pain 7-9: severe pain 10: worst pain imaginable

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Forces Institute of dentistry, Rawalpindi, Punjab Province, Pakistan